CLINICAL TRIAL: NCT01062087
Title: Retrospective Investigation of Postoperative Pain Perception After Laparoscopic Tubal Sterilization
Brief Title: Pain Perception After Tubal Ligation
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Principal Investigator, Sarah McCoy, OB/GYN, Oklahoma State University Center for Health Sciences
Other Study IDs: 2010002
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: postoperative pain; tubal ligation; local anesthetic
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Local anesthetic: Women who received local anesthetic during surgery in addition to general anesthesia
  Interventions: Drug: Bupivacaine, Lidocaine
- No local anesthetic: Women who did not receive any local anesthetic during surgery, but did have general anesthesia

INTERVENTIONS:
Drug: Bupivacaine, Lidocaine — Injection at surgical port site of 0.25% Bupivicaine, 2.5 mg/mL NaCl solution and/or application of Lidocaine HCl jelly 2% aqueous, up to 5 mL
  Other Names: Marcaine
  Groups: Local anesthetic

SUMMARY:
The purpose of this study is to attempt to determine retrospectively whether there was a statistically significant difference in patient need for postoperative narcotics between two different groups of women who received a laparoscopic tubal ligation. One group received a local anesthetic injection or gel at the surgical sites, in addition to general anesthesia. The other group did not receive any local anesthetic but did receive general anesthesia. The investigators hypothesize that the group that received the local anesthetic injection or gel had lower average postoperative narcotic requirements and shorter postoperative dismissal to home times than the group that did not receive the auxiliary local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 21-52,having a laparoscopic tubal ligation by the fallopia ring method at Oklahoma State University Medical Center between January 1, 2005 and December 31, 2009

Exclusion Criteria:

* We will exclude women with the following comorbid conditions, since they may alter the patient's pain level or her perception of pain after the tubal ligation: history of chronic pelvic pain, history of pelvic inflammatory disease, opiate abuse, conversion to open procedure, unsuccessful tubal ligation, laceration of tube, more than one ring placed on single tube, admittance to the hospital, additional procedures performed, endometriosis, allergy to marcaine, lidocaine, or bupivicaine.

Ages: 21 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Urban clinic population, mix of ethnicities, most are Medicaid patients
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Amount of postoperative narcotic required before dismissal from hospital | up to 12 hours

SECONDARY OUTCOMES:
The amount of time required for postoperative hospitalization before dismissal | 2-12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Terry Badzinski, DO, Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- Oklahoma State University Medical Center, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Bordahl PE, Raeder JC, Nordentoft J, Kirste U, Refsdal A. Laparoscopic sterilization under local or general anesthesia? A randomized study. Obstet Gynecol. 1993 Jan;81(1):137-41. PMID 8416449
- [Background] Benhamou D, Narchi P, Mazoit JX, Fernandez H. Postoperative pain after local anesthetics for laparoscopic sterilization. Obstet Gynecol. 1994 Nov;84(5):877-80. PMID 7936530